CLINICAL TRIAL: NCT00328159
Title: Dietary Therapy of Mitochondrial Fatty Acids Oxidation. A Clinical Study of Treatment With Odd Carbons Medium-chain Fatty Acids
Brief Title: Nutritional Therapy of the Deficits of Oxidation Mitochondrial of the Fatty Acids
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Marie CASTERA, Department of Clinical Research of developpement
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: P030435
Record Dates: First submitted 2006-05-18; First posted 2006-05-19 (Estimated); Last update posted 2011-02-17 (Estimated); Status verified 2007-03

CONDITIONS: Inborn Errors of Metabolism
Keywords: FAO disorders; long-chain FAO enzyme defects; inborn errors of metabolism; carnitine palmitoyltransferase 1 (CPT1),; carnitine-acylcarnitine translocase (CAT),; carnitine palmitoyltransferase 2 (CPT2),; very-long chain acyl-CoA dehydrogenase (VLCAD),; L-3-hydroxy-acyl-CoA dehydrogenase (LCHAD); or trifunctional protein (MTP).
MeSH Terms: conditions — Metabolism, Inborn Errors; VLCAD deficiency

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Oil special 107 and MYGLIOL 810

SUMMARY:
Usual dietary therapies of mitochondrial fatty acid oxidation disorders (FAO) are based on 3 strategies:

* limitation of lipid intake in the diet;
* supplementation of the diet with medium-chain triglycerides (MCT) for patients affected with disorders of long-chain FAO;
* some specific supplementations (for example, L-carnitine).

These strategies are often ineffective. The aim of the present study is to evaluate new therapeutic ways based on the underlying energetic defect observed in these disorders. The long-term goal is to develop efficient therapies of these disorders.

DETAILED DESCRIPTION:
The main specific aim of this study will be to determine the efficiency of odd-chain MCT: TRIHEPTANOIN (Tri-C7) and its metabolites, BETA-HYDROXYPENTANOATE (BHP) and BETA-KETOPENTANOATE (BKP), as potential treatments by orale or enteral routes. These compounds are efficiently used for energy production, despite long-chain FAO enzyme defects. They use alternative metabolic pathways and have anaplerotic effects due to propionyl-CoA production by the thiolytic cleavage of odd carbon ketone bodies.

The efficiency of these compounds will be compared with conventional diet (MCT) for each patient. Because of frequent phenotypic variations observed for each of these diseases, each patient will be his own control.

The same protocol study will be followed in 2 centers: Dallas, USA (main investigator: Dr CR Roe) and Paris, France (main investigator: Dr G TOUATI). It is planned to include 80 patients (60 in Dallas, 20 in Paris), during the next 2 years. The patients will be affected with 6 proven defects that are specific defects of long-chain FAO: carnitine palmitoyltransferase 1 (CPT1), carnitine-acylcarnitine translocase (CAT), carnitine palmitoyltransferase 2 (CPT2), very-long chain acyl-CoA dehydrogenase (VLCAD), L-3-hydroxy-acyl-CoA dehydrogenase (LCHAD) or trifunctional protein (MTP).

The used methodology will be a control randomized study to compare the efficiency of 2 diet therapies: TRIHEPTANOIN versus conventional MCT. The studied parameters will depend on each disease and will depend on the affected organs in each patient. Main studied clinical parameters will be: survival rate, number of metabolic acute decompensation, frequency and severity of hypoglycemias, frequency and severity of rhabdomyolyses, evolution of cardiac or hepatic manifestations, muscular strength, and quality of life. Main studied biological parameters will be: TRIHEPTANOIN use during meal tests, modifications of plasma acylcarnitines profile, modifications of urinary organic acids, blood measurements of CPK and transaminases. Cardiac echographies will be performed for the follow-up of cardiomyopathies, ergometric testing and strength tests will be performed for disorders that affect muscular function.

ELIGIBILITY:
Inclusion Criteria:

* Patient with an enzyme deficiency of carnitine palmitoyltransferase 1 (CPT1), carnitine-acylcarnitine translocase (CAT), carnitine palmitoyltransferase 2 (CPT2), very-long chain acyl-CoA dehydrogenase (VLCAD), L-3-hydroxy-acyl-CoA dehydrogenase (LCHAD) or trifunctional protein (MTP).
* Covered by health and social insurance
* Written informed consent

Exclusion Criteria:

* Patient affected with FAO dysfunction secondary to other cause (e.g. mitochondrial respiratory chain disorders)
* Patient with suspected FAO disorder that has not been proven (by enzymatic or molecular test)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2006-06; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
Strength tests | 24 months
Biological parameters (acylcarnitines profile, modifications of urinary organic acids) | 24 months
Clinical parameters (echocardiography) | 24 months

SECONDARY OUTCOMES:
Ergometric testing | 24 months
Hepatic functions | 24 months
Hypoglycaemia | 24 months
Rhabdomyolyses | 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Guy Touati, PU-PH, Principal Investigator — Assistance Publique Hopitaux de Paris
Locations (1):
- Necker University Hospital - Metabolism Unit, Paris, France